CLINICAL TRIAL: NCT05593965
Title: Causal Role of Frontostriatal Circuitry in Goal-directed Behavior
Acronym: NANCY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 22-2430; 1K99MH126161-01A1 (NIH)
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Results first posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2023-09

CONDITIONS: Executive Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- TMS to lateral prefrontal cortex followed by TMS to medial prefrontal cortex (Experimental): Participants will receive TMS while performing a reward-based decision-making task. In the first stimulation session, the TMS coil will be placed over the lateral prefrontal cortex on the scalp. In the second session, the TMS coil will be placed over the medial prefrontal cortex on the scalp. during every session, subjects receive Delta-beta patterned TMS, Theta-gamma patterned TMS, and Arrhythmic TMS.
  Interventions: Device: Delta-beta TMS; Device: Theta-gamma TMS; Device: Arrhythmic TMS
- TMS to medial prefrontal cortex followed by TMS to lateral prefrontal cortex (Experimental): Participants will receive TMS while performing a reward-based decision-making task. In the first stimulation session, the TMS coil will be placed over the medial prefrontal cortex on the scalp. In the second session, the TMS coil will be placed over the lateral prefrontal cortex on the scalp. during every session, subjects receive Delta-beta patterned TMS, Theta-gamma patterned TMS, and Arrhythmic TMS.
  Interventions: Device: Delta-beta TMS; Device: Theta-gamma TMS; Device: Arrhythmic TMS

INTERVENTIONS:
Device: Delta-beta TMS — TMS will be delivered in a delta-beta pattern in which triplets of pulses delivered at 20 Hz (50 milliseconds between each pulse) are sent every 3 Hz (333 milliseconds between the start of each triplet).
Device: Theta-gamma TMS — TMS will be delivered in a theta-gamma pattern in which triplets of pulses delivered at 50 Hz (20 milliseconds between each pulse) are sent every 5 Hz (200 milliseconds between the start of each triplet).
Device: Arrhythmic TMS — TMS will be delivered in an arrhythmic pattern in which pulses are delivered with a random inter-pulse interval. The number of pulses and duration is matched to that of the Delta-beta TMS and Theta-gamma TMS.

SUMMARY:
The purpose of this clinical trial is to investigate the causal role that frontostriatal circuitry plays in goal-directed behavior. The participants will perform a reward-based decision-making task. During the task, cross-frequency patterned rhythmic transcranial magnetic stimulation (TMS) will be delivered at delta-beta frequency, a control-frequency, or an active sham to either the dorsolateral or medial prefrontal cortex (PFC). Electroencephalography will be collected concurrent with stimulation. Structural and functional magnetic resonance imaging (MRI) will be collected during performance of the reward-based decision-making task to localize the stimulation targets.

DETAILED DESCRIPTION:
This study is a pilot, four-session, crossover study with transcranial magnetic stimulation (TMS), electroencephalography (EEG), and magnetic resonance imaging (MRI) to understand the causal role of delta-beta coupling in goal-directed behavior in the dorsolateral prefrontal cortex (dlPFC) to dorsal striatum circuit. Participants that request to be in the experiment will provide verbal, documented consent to undergo a phone screening to assess that the participant meets initial exclusion/inclusion criteria. Participants complete an MRI and TMS screening form over the phone to ensure eligibility.

The first session will be an EEG session with the reward-based decision-making task. At the start of the session, the investigators will acquire written informed consent. Then, the investigators will administer a pregnancy test if applicable. Participants will complete five assessments: the Snaith Hamilton Pleasure Scale, Behavioral Activation System and Behavioral Inhibition System, Temporal Experience of Pleasure Scale, the State-Trait Anxiety Inventory, and Ruminative Responses Scale. Note that the participants are from a convenient sample and are not required to be diagnosed with major depressive disorder. Thus, these assessments were selected as they survey various personality traits that might be relevant to performance in the task.

The scalp dimensions of each participant are calculated and an EEG net is applied. Next, the participants complete an eyes-open and eyes-closed resting-state recording of EEG. Then, the streamlined version of the Expenditure of Effort for Reward Task (S-EEfRT) is completed. These data serve as baseline measurement of brain activity without any form of stimulation. This session takes approximately 1.5 hours to complete. After each block of the task, the task difficulty will increase or decrease based on performance. At the end of the session, if the participant chose to perform the hard task greater than 85% of the time or less than 15% of the time, then the participant will not be invited to the next session of the experiment. Participants that do not dynamically change their response based on the incentive are not engaged with the relevant cognitive constructs under investigation in this study.

The second session takes place at the MRI facility. In the 24 hours prior to this session, participants complete an MRI screening form to ensure eligibility based on common contraindications for MRI. During the 60 minutes of scanning, a 5-minute structural MR is acquired and the remaining time is used to complete as many blocks of the S-EEfRT as possible. The minimal number of sessions required to use the data is 5 blocks, which requires approximately 25 minutes to collect. If a participant was unable to complete the requisite number of sessions, then they will be excluded from the study. Functional MRI data is analyzed before the 3rd and 4th session to localize the regions of dorsolateral prefrontal cortex (dlPFC) and medial prefrontal cortex (mPFC) for stimulation. In the localization analysis, a region of interest mask in the head of the left caudate and in left nucleus accumbens are drawn and the region in dlPFC and mPFC with peak functional connectivity in task-based functional connectivity to these regions. In a pilot dataset collected by the investigators, it was found that the contrast of trails in which there was a decision to perform the hard task versus trials in which the easy task was selected was sufficient to localize the anterior middle frontal gyrus. The contrast of trials in which high versus low incentive was offered was sufficient to localize the medial prefrontal cortex. Thus, the investigators will choose regions in these anatomical areas with maximal connectivity to their respective nucleus in the striatum.

The order of regions (dlPFC then mPFC, or mPFC then dlPFC) targeted by TMS in the third and fourth session will be randomized and counter-balanced. In the third and fourth session, participants will complete a TMS contraindications screening form. The same TMS screening form will be administered over the phone and at the start of each of the TMS session. If there is any ambiguity in the contraindications for the TMS form, then the medical monitor who is an epileptologist is consulted and final approval is acquired. Participants will be fitted with a low-profile EEG net. In the third session, the motor threshold of each participant will be calculated using single-pulse TMS to the hand knob of the left primary motor cortex with real-time monitoring of the motor-evoked potential using electrodes on the first dorsal interosseus muscle. Researchers may also use visible twitch to calculate the motor threshold. The motor threshold is defined as the percent stimulator output when a motor-evoked potential or visible twitch is observed approximately 50% of the time. For the fourth session, the same stimulator intensity will be used as in the third session. The structural MRI and regions of interest (dlPFC and mPFC) are imported into neuronavigation software. The participant wears a three-dimensional stereotaxic tracking headband and their head is registered to their structural MRI using canonical coordinates on the scalp. Then, the TMS coil is targeted to either mPFC or dlPFC and the position of the coil relative to the head is recorded throughout the session. The participant performs the S-EEfRT as the patterned trains of TMS are delivered on every trial. Each block of the study is randomized to receive either delta-beta patterned (triplets of TMS pulses at 20 Hertz every 3 Hertz), theta-gamma patterned (triplets of pulses at 50 Hertz every 5 Hertz), or an arrhythmic pattern (same number of pulses and duration with a random inter-pulse interval). After stimulation, a questionnaire is provided with common side effects of TMS. Based on the results of the stimulation side effects questionnaire, a structured adverse events interview is conducted to acquire more information regarding any side effects that were selected to be "very high" by the participant. The third and fourth session will each take approximately two hours.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Between the ages of 18 and 35
* Right handed
* Able to provide informed consent
* Willing to comply with all study procedures
* Available for the duration of the study
* Speak and understand English.

Exclusion Criteria:

* Attention Deficit Hyperactivity Disorder (currently under treatment)
* Neurological disorders and conditions, including, but not limited to: History of epilepsy Seizures (except childhood febrile seizures)
* Dementia
* History of stroke
* Parkinson's disease
* Multiple sclerosis
* Cerebral aneurysm
* Brain tumors
* Medical or neurological illness or treatment for a medical disorder that could interfere with study participation (e.g., unstable cardiac disease, human immunodeficiency virus or acquired immunodeficiency syndrome, malignancy, liver or renal impairment)
* Prior brain surgery
* Any brain devices/implants, including cochlear implants and aneurysm clips
* Cardiac pacemaker
* Any other implanted electronic device
* History of current traumatic brain injury
* (For females) Pregnancy or breast feeding
* Anything that, in the opinion of the investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board, Independent Ethics Committee, or Research Ethics Board, as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Starting 9 months and continuing for 36 months following publication
Access Criteria: Deidentified individual data that supports the results will be shared provided the investigator who proposes to use the data has approval from an Institutional Review Board, Independent Ethics Committee, or Research Ethics Board and an executed data use/sharing agreement with the University of North Carolina at Chapel Hill.

RESULTS

PARTICIPANT FLOW:
Groups:
- TMS to Lateral Prefrontal Cortex Followed by TMS to Medial Prefrontal Cortex: Participants will receive transcranial magnetic stimulation (TMS) while performing a reward-based decision-making task. In the first stimulation session, the TMS coil will be placed over the lateral prefrontal cortex on the scalp. In the second session, the TMS coil will be placed over the medial prefrontal cortex on the scalp. during every session, subjects receive Delta-beta patterned TMS, Theta-gamma patterned TMS, and Arrhythmic TMS.
  Delta-beta TMS: TMS will be delivered in a delta-beta pattern in which triplets of pulses delivered at 20 Hz (50 milliseconds between each pulse) are sent every 3 Hz (333 milliseconds between the start of each triplet).
  Theta-gamma TMS: TMS will be delivered in a theta-gamma pattern in which triplets of pulses delivered at 50 Hz (20 milliseconds between each pulse) are sent every 5 Hz (200 milliseconds between the start of each triplet).
  Arrhythmic TMS: TMS will be delivered in an arrhythmic pattern in which pulses are delivered with a random inter-pulse interval. The number of pulses and duration is matched to that of the Delta-beta TMS and Theta-gamma TMS.
Period: 1st Intervention (1 Day)
Arm/Group | TMS to Lateral Prefrontal Cortex Followed by TMS to Medial Prefrontal Cortex | TMS to Medial Prefrontal Cortex Followed by TMS to Lateral Prefrontal Cortex
Started | 17 | 7
Completed | 16 | 7
Not Completed | 1 | 0
Not completed — Technical error | 1 | 0
Period: 2nd Intervention (1 Day)
Arm/Group | TMS to Lateral Prefrontal Cortex Followed by TMS to Medial Prefrontal Cortex | TMS to Medial Prefrontal Cortex Followed by TMS to Lateral Prefrontal Cortex
Started | 16 | 7
Completed | 16 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TMS to Lateral Prefrontal Cortex Followed by TMS to Medial Prefrontal Cortex | TMS to Medial Prefrontal Cortex Followed by TMS to Lateral Prefrontal Cortex | Total
Number analyzed (Participants) | 17 | 7 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 7 | 24
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.4 (4.4) | 23.3 (6.0) | 22.0 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 5 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 7 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 2 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 8 | 4 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 7 | 24
Percentage of the Trials That the Participant Chooses to Perform the Hard Task [Mean (Standard Deviation); unit: percentage of trials] — In the Expenditure of Effort for Reward Task, participants are faced with a decision on every trial: to choose an easy task with a low effort exertion for a chance at winning a low amount of money and a hard task with a high effort exertion for a chance at winning a greater amount of money. The incentive for the high effort exertion is changed on each trial and the participant gets physically tired from repeated effort exertion. Goal-directed behavior was calculated as the percentage of trials in which the participant decides to perform the most difficult effort exertion task in the task.
  percentage of trials | 54.0 (12.8) | 56.9 (11.2) | 54.8 (12.2)
Coupling Strength Between Low-frequency Prefrontal Signals and High-frequency Posterior Signals [Mean (Standard Deviation); unit: Z-score] — Phase-amplitude coupling strength is calculated using the mean vector length metric between low-frequency activity in prefrontal electrodes and high-frequency activity in motor electrodes. A Z-score indicates the number of standard deviations away from the mean of distribution generated by randomly time-shifting the data. A Z-score of 0 is equal to the mean coupling strength of random data. Higher values are greater coupling strength. Positive values (> 1) indicate increased prefrontal control over the motor cortex, which is found in healthy individuals during decision-making.
  Z-score | 0.414 (1.071) | -0.179 (1.401) | 0.345 (1.106)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of the Trials That the Participant Chooses to Perform the Hard Task
Description: In the Expenditure of Effort for Reward Task, participants are faced with a decision on every trial: to choose an easy task with a low effort exertion for a chance at winning a low amount of money and a hard task with a high effort exertion for a chance at winning a greater amount of money. The incentive for the high effort exertion is changed on each trial and the participant gets physically tired from repeated effort exertion. Goal-directed behavior was calculated as the percentage of trials in which the participant decides to perform the most difficult effort exertion task in the Expenditure of Effort for Reward Task. A higher percentage equates to more goal-directed behavior and is favorable.
Time Frame: 2 hours during the 1st intervention and 2 hours during the 2nd intervention
Measure: Mean (Standard Deviation); unit: Percentage of trials
Groups:
- Delta-beta TMS to Lateral Prefrontal Cortex: Participants received delta-beta TMS to lateral prefrontal cortex while performing a reward-based decision-making task. Delta-beta TMS: TMS will be delivered in a delta-beta pattern in which triplets of pulses delivered at 20 Hz (50 milliseconds between each pulse) are sent every 3 Hz (333 milliseconds between the start of each triplet).
- Theta-gamma TMS to Lateral Prefrontal Cortex: Participants received theta-gamma TMS to lateral prefrontal cortex while performing a reward-based decision-making task. Theta-gamma TMS: TMS will be delivered in a theta-gamma pattern in which triplets of pulses delivered at 50 Hz (20 milliseconds between each pulse) are sent every 5 Hz (200 milliseconds between the start of each triplet).
- Arrhythmic TMS to Lateral Prefrontal Cortex: Participants received arrhythmic TMS to lateral prefrontal cortex while performing a reward-based decision-making task. Arrhythmic TMS: TMS will be delivered in an arrhythmic pattern in which pulses are delivered with a random inter-pulse interval. The number of pulses and duration is matched to that of the Delta-beta TMS and Theta-gamma TMS.
- Delta-beta TMS to Medial Prefrontal Cortex: Participants received delta-beta TMS to medial prefrontal cortex while performing a reward-based decision-making task. Delta-beta TMS: TMS will be delivered in a delta-beta pattern in which triplets of pulses delivered at 20 Hz (50 milliseconds between each pulse) are sent every 3 Hz (333 milliseconds between the start of each triplet).
- Theta-gamma TMS to Medial Prefrontal Cortex: Participants received theta-gamma TMS to medial prefrontal cortex while performing a reward-based decision-making task. Theta-gamma TMS: TMS will be delivered in a theta-gamma pattern in which triplets of pulses delivered at 50 Hz (20 milliseconds between each pulse) are sent every 5 Hz (200 milliseconds between the start of each triplet).
- Arrhythmic TMS to Medial Prefrontal Cortex: Participants received arrhythmic TMS to medial prefrontal cortex while performing a reward-based decision-making task. Arrhythmic TMS: TMS will be delivered in an arrhythmic pattern in which pulses are delivered with a random inter-pulse interval. The number of pulses and duration is matched to that of the Delta-beta TMS and Theta-gamma TMS.
Arm/Group | Delta-beta TMS to Lateral Prefrontal Cortex | Theta-gamma TMS to Lateral Prefrontal Cortex | Arrhythmic TMS to Lateral Prefrontal Cortex | Delta-beta TMS to Medial Prefrontal Cortex | Theta-gamma TMS to Medial Prefrontal Cortex | Arrhythmic TMS to Medial Prefrontal Cortex
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 23 | 23
Percentage of trials | 33.2 (22.2) | 32.9 (20.1) | 33.6 (21.0) | 37.1 (21.6) | 37.1 (21.9) | 37.6 (19.5)

2. Secondary Outcome: Coupling Strength Between Low-frequency Prefrontal Signals and High-frequency Posterior Signals
Description: Phase-amplitude coupling strength is calculated using the mean vector length metric between low-frequency activity in prefrontal electrodes and high-frequency activity in motor electrodes. A Z-score indicates the number of standard deviations away from the mean of distribution generated by randomly time-shifting the data. A Z-score of 0 is equal to the mean coupling strength of random data. Higher values are greater coupling strength. Positive values (> 1) indicate increased prefrontal control over the motor cortex, which is found in healthy individuals during decision-making.
Time Frame: 2 hours during the 1st intervention and 2 hours during the 2nd intervention
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Delta-beta TMS to Lateral Prefrontal Cortex | Theta-gamma TMS to Lateral Prefrontal Cortex | Arrhythmic TMS to Lateral Prefrontal Cortex | Delta-beta TMS to Medial Prefrontal Cortex | Theta-gamma TMS to Medial Prefrontal Cortex | Arrhythmic TMS to Medial Prefrontal Cortex
Number analyzed (Participants) | 23 | 23 | 23 | 23 | 23 | 23
Z-score | 0.416 (1.073) | 0.008 (1.214) | 0.308 (1.112) | -0.051 (1.241) | -0.094 (0.850) | 0.274 (1.027)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored during the first and second intervention, a total of four hours across 1 week
Description: In this cross-over design, the interventions were administered in a block design such that each block included the same type of stimulation (delta-beta, theta-gamma, or arrhythmic patterned). Adverse events were assessed at the end of the session. Thus, there are adverse events reported for each stimulation location (lateral prefrontal cortex or medial prefrontal cortex), but there is no way to determine which of the patterns of stimulation might be more or less related to the adverse events.
Groups:
- TMS to Lateral Prefrontal Cortex: Participants received TMS to the lateral prefrontal cortex while performing a reward-based decision-making task.
- TMS to Medial Prefrontal Cortex: Participants received TMS to the medial prefrontal cortex while performing a reward-based decision-making task.
Arm/Group | TMS to Lateral Prefrontal Cortex | TMS to Medial Prefrontal Cortex
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 1/24 | 0/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMS to Lateral Prefrontal Cortex (N=24) | TMS to Medial Prefrontal Cortex (N=23)
Trouble concentrating (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT05593965/Prot_SAP_001.pdf
  • Informed Consent Form (2022-12-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT05593965/ICF_000.pdf